CLINICAL TRIAL: NCT05339087
Title: Efficacy and Safety of Riociguat (MK-4836) in Incipient Pulmonary Vascular Disease as an Indicator for Early Pulmonary Arterial Hypertension Double-blind, Randomized, Multicenter, Multinational, Placebo-controlled Phase IIa Study (ESRA)
Brief Title: Efficacy and Safety of Riociguat in Incipient Pulmonary Vascular Disease as an Indicator for Early PAH
Acronym: ESRA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Strategic re-prioritization by the IMP supplier. Decision not safety-related.
Sponsor: Heidelberg University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Prof. Dr. med. Ekkehard Gruenig, Head of section for pulmonary hypertension, Thoraxklinik Heidelberg gGmbH, Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-01RCT
Record Dates: First submitted 2022-04-14; First posted 2022-04-21 (Actual); Results first posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Pulmonary Vascular Disorder; Primary Pulmonary Hypertension; Systemic Sclerosis; Other Systemic Involvement of Connective Tissue
Keywords: early pulmonary vascular disease; riociguat; pulmonary hypertension
MeSH Terms: conditions — Familial Primary Pulmonary Hypertension; Scleroderma, Systemic; Hypertension, Pulmonary | interventions — riociguat

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Riociguat (Experimental): patients will undergo a titration phase starting with 1mg riociguat oral tablets tid (three times daily) up to a maximum dosage of 2.5mg tid that will be continued for the remainder of the study.
  Interventions: Drug: Riociguat Oral Tablet
- Placebo (Placebo Comparator): Placebo tablets with the same treatment regimen (tid) as the verum therapy will be provided. Patients will undergo a sham titration phase with sham doses individually adjusted as in the experimental arm
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Riociguat Oral Tablet — Riociguat Oral Tablet (1 mg, 1.5 mg, 2.0 mg or 2.5 mg three times daily) Titration phase: dose will be individually adjusted in accordance with the in-label titration regimen. Dose adjustment will be performed every two weeks by phone taking the systemic blood pressure of the patient, the subjects and physicians' subjective estimation and occurrence of adverse reactions into account. At week 8 the maintenance dose will be established and continued for the rest of the study
  Other Names: MK-4836; ATC Code: C02KX05
  Arms: Riociguat
Other: Placebo — Sham titration and adjustment to maintenance dose will be performed according to individual tolerability as in the experimental arm.
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, multicenter, multinational study investigating the effect of riociguat (MK-4836) in patients with early pulmonary vascular disease.

DETAILED DESCRIPTION:
Chronic pulmonary arterial hypertension (PAH) is associated with impaired exercise capacity, quality of life and right ventricular function characterized by an increase of pulmonary vascular resistance (PVR) and pulmonary arterial pressure, leading to right heart insufficiency.

Riociguat tratment is approved for both PAH and chronic thromboembolic pulmonary hypertension (CTEPH).

Data on early treatment of patients with mildly elevated pulmonary arterial pressures is still scarce but there is evindence that such patients may benefit from early targeted therapy.

For instance, in a trial on systemic sclerosis (SSc)-patients with mildly elevated mean pulmonary artery pressure (mPAP) and/or exercise pulmonary hypertension, without significant left heart or lung disease, ambrisentan, an endothelin receptor antagonist resulted in an improvement of PVR as secondary endpoint, which may be of prognostic relevance in this patient cohort and requires further research.

Besides its prognostic significance among patients with SSc-APAH, PVR may be an indicator of early pulmonary vascular disease and previous studies proved the positive effects of riociguat on right heart size and PVR (secondary endpoint in phase III studies). Thus, PVR was chosen as primary endpoint of this study aiming to investigate the effect of riociguat (MK-4836) on PVR, clinical parameters, safety and tolerability in patients with early pulmonary vascular disease.

Eligible subjects will be randomized in a 1:1 ratio to receive either riociguat or placebo.

Medical examinations include medical history, physical examination, electrocardiogram, blood gas analyses, lung function tests, laboratory testing (including NT-proBNP), echocardiography at rest, and right heart catheterization.

The prospective period of data collection comprises a 24-week treatment phase diveded into an 8-week titration phase followed by a 16-week main study phase as well as a safety follow-up of 30±14 days.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age at time of inclusion.
2. Male and female patients with early pulmonary vascular disease, defined as either a) mean pulmonary arterial pressure (mPAP) ≥25 mmHg with pulmonary vascular resistance (PVR) ≥2 to <3 WU and pulmonary arterial wedge pressure (PAWP) ≤15 mmHg or b) mPAP 21-<25 mmHg with PVR ≥2 WU, and PAWP ≤15 mmHg associated with connective tissue disease (CTD) or as idiopathic/heritable form (see Group I / Nice Clinical Classification of Pulmonary Hypertension) (acc. to Simonneau et al. 2019). Patients with rheumatoid arthritis or connective tissue disease of any kind, except systemic lupus erythematosus, may also be included. Patients in group b will be mainly enrolled as long as patients in group a are not defined as having pulmonary arterial hypertension according to European pulmonary hypertension guidelines.
3. Treatment naïve patients (with respect to PAH specific medication)
4. Unspecific treatments which may also be used for the treatment of pulmonary hypertension such as oral anticoagulants, diuretics, digitalis, calcium channel blockers or oxygen supplementation are permitted. Permitted are also treatments of the rheumatologic disease. However, these drugs must have been started at least 1 month before right heart catheterization.
5. Right-heart catheterization results must not be older than 1 month at Visit 1 (will be considered as baseline values, the time frame can be prolonged up to 6 months, if the patient has had no signs of clinical changes defined as >10% change of 6MWD, WHO FC, > 30% change in NT-proBNP) and must have been measured in the participating center under standardized conditions (refer to the study specific Swan Ganz catheterization manual). If the respective measurements have not been performed in context with the patient's regular diagnostic work up, they have to be performed as a part of the study during the pre-study phase (after the patient signed the informed consent).
6. Women without childbearing potential defined as postmenopausal women aged 55 years or older, women with bilateral tubal ligation, women with bilateral ovariectomy, and women with hysterectomy can be included in the study.
7. Women of childbearing potential can only be included in the study if all of the following applies (listed below):

   1. Negative serum pregnancy test at screening and at study start (visit 1).
   2. Agreement to undertake monthly urine pregnancy tests during the study and up to at least 30 days after study treatment discontinuation. These tests should be performed by the patient at home.
   3. Agreement to use a highly effective contraception method as specified from screening until at least 30 days after last dose of study medication.
8. Patients who are able to understand and follow instructions and who are able to participate in the study for the entire period.
9. Patients must have given their written informed consent to participate in the study after having received adequate previous information and prior to any study-specific procedures.

Exclusion Criteria:

1. Patients with systemic lupus erythematosus.
2. Concomitant PAH-targeted treatment is not allowed during the study.
3. Concomitant treatment with phosphodiesterase 5 inhibitors, endothelin receptor antagonists and prostacyclin analogues due to digital ulcers is contraindicated and must not be taken during the study period. Such drugs must have a washout-phase of 3 days at the time of right heart catheterization at screening. Intravenous treatment with prostacyclin analogues should not be performed within 1 week of right heart catheterization. Any decision to discontinue above-mentioned drugs will be made by the clinicians and the patient at screening, which takes part during the patients' regular routine visit. The discontinuation of above-mentioned drugs will be evaluated by considering the presence or absence of digital ulcers and their frequency of appearance in the patient's medical history.
4. Pulmonary hypertension explained by other cause including group 2, 3, 4 and 5 PH according to the current guidelines.
5. Cardiac comorbidity, defined with three or more of the following conditions: uncontrolled arterial hypertension, diabetes mellitus, body mass index >35, left atrial enlargement >20 cm², atrial fibrillation, left ventricular ejection fraction <50%.
6. Pulmonary comorbidity, defined as forced vital capacity (FVC) ≤70; forced expiratory volume in 1 second (FEV1) ≤50%; diffusion capacity of the lung (DLCO) ≤40%. FVC may be <70/ if high resolution computed tomography shows <20% lung fibrosis.
7. Patients with a medical disorder, condition, or history of such that would impair the patient's ability to participate or complete this study in the opinion of the investigator.
8. Patients with underlying medical disorders with an anticipated life expectancy below 2 years (e.g. active cancer disease with localized and/or metastasized tumor mass).
9. Patients with a history of severe or multiple drug allergies (defined as allergic reactions to three or more structurally unrelated drugs).
10. Patients with hypersensitivity to the investigational drug or any of the excipients.
11. Contraindications according to summary of product characteristics of riociguat (e.g. arterial hypotension with systolic blood pressure <95 mmHg; nitrates)
12. Participation in any clinical drug trial within 4 weeks prior to screening of this study and/or patient, who is scheduled to receive an investigational medicinal product (IMP) during the course of this study
13. Background therapy with highly anti-fibrotic drugs (pirfenidone) or nintedanib, prednisolone >10 mg/day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-10-24 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ekkehard Grünig, MD, Principal Investigator — Thoraxklinik at the University of Heidelberg
Locations (8):
- Austria (2):
  - LKH-Univ. Klinikum Graz Universitätsklinik für Innere Medizin Klinische Abteilung für Pulmonologie, Graz
  - Ordensklinikum Linz GmbH Elisabethinen, Linz
- Centre de référence des Maladies Auto-Immunes Systémiques rares du Nord et Nord-Ouest (CeRAINO) Service de Médecine Interne et Immunologie Clinique Hôpital Claude Huriez, CHU, Lille, France
- Germany (2):
  - Carl Gustav Carus University Hospital at the TU Dresden, Medical Department I, Center for PH, Dresden
  - Centre for Pulmonary Hypertension at the Thoraxklinik Heidelberg, Heidelberg University Hospital Heidelberg, Heidelberg
- Università Degli Studi Di Napoli Federico II Scuola Di Medicina E Chirurgia, Napoli, Italy
- Universitätsspital Zürich Pulmonale Hypertonie, Klinik für Pneumologie, Zurich, Switzerland
- Royal Free London NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Galie N, Humbert M, Vachiery JL, Gibbs S, Lang I, Torbicki A, Simonneau G, Peacock A, Vonk Noordegraaf A, Beghetti M, Ghofrani A, Gomez Sanchez MA, Hansmann G, Klepetko W, Lancellotti P, Matucci M, McDonagh T, Pierard LA, Trindade PT, Zompatori M, Hoeper M. 2015 ESC/ERS Guidelines for the Diagnosis and Treatment of Pulmonary Hypertension. Rev Esp Cardiol (Engl Ed). 2016 Feb;69(2):177. doi: 10.1016/j.rec.2016.01.002. No abstract available. PMID 26837729
- [Background] Grunig E, Barner A, Bell M, Claussen M, Dandel M, Dumitrescu D, Gorenflo M, Holt S, Kovacs G, Ley S, Meyer JF, Pabst S, Riemekasten G, Saur J, Schwaiblmair M, Seck C, Sinn L, Sorichter S, Winkler J, Leuchte HH. [Non-invasive diagnosis of pulmonary hypertension: ESC/ERS Guidelines with commentary of the Cologne Consensus Conference 2010]. Dtsch Med Wochenschr. 2010 Oct;135 Suppl 3:S67-77. doi: 10.1055/s-0030-1263314. Epub 2010 Sep 22. German. PMID 20862623
- [Background] Ghofrani HA, D'Armini AM, Grimminger F, Hoeper MM, Jansa P, Kim NH, Mayer E, Simonneau G, Wilkins MR, Fritsch A, Neuser D, Weimann G, Wang C; CHEST-1 Study Group. Riociguat for the treatment of chronic thromboembolic pulmonary hypertension. N Engl J Med. 2013 Jul 25;369(4):319-29. doi: 10.1056/NEJMoa1209657. PMID 23883377
- [Background] Pan Z, Marra AM, Benjamin N, Eichstaedt CA, Blank N, Bossone E, Cittadini A, Coghlan G, Denton CP, Distler O, Egenlauf B, Fischer C, Harutyunova S, Xanthouli P, Lorenz HM, Grunig E. Early treatment with ambrisentan of mildly elevated mean pulmonary arterial pressure associated with systemic sclerosis: a randomized, controlled, double-blind, parallel group study (EDITA study). Arthritis Res Ther. 2019 Oct 26;21(1):217. doi: 10.1186/s13075-019-1981-0. PMID 31655622
- [Background] Rubin LJ, Galie N, Grimminger F, Grunig E, Humbert M, Jing ZC, Keogh A, Langleben D, Fritsch A, Menezes F, Davie N, Ghofrani HA. Riociguat for the treatment of pulmonary arterial hypertension: a long-term extension study (PATENT-2). Eur Respir J. 2015 May;45(5):1303-13. doi: 10.1183/09031936.00090614. Epub 2015 Jan 22. PMID 25614164

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at 6 study centres between October 2022 and May 2025. The first participant was enrolled on 24 October 2022, the last on 30 May 2025.
Pre-assignment Details: Overall, 35 participants met the eligibility criteria and were randomized to treatment.
Groups:
- Riociguat: Riociguat oral tablet (1 mg, 1.5 mg, 2.0 mg or 2.5 mg three times daily): individually adjusted dose in accordance with the in-label titration regimen (maximum dosage of 2.5mg tid). At week 8, the maintenance dose was established and maintained for the rest of study participation.
- Placebo: Placebo oral tablets: Sham titration and adjustment to maintenance dose (tid) according to individual tolerability as in the experimental arm.
Period: Overall Study
Arm/Group | Riociguat | Placebo
Started | 17 | 18
Visit 2 | 13 (Skipped visit 2 (n = 3): Early study termination (n = 1); Early termination of trial medication (n = 1); own request (n = 1)) | 14 (Skipped visit 2 (n = 3) Early study termination (n = 2) Early termination of trial medication (n = 1))
Visit 3 | 16 (Premature visit 3 (n = 4 out of 16): Early study termination (n = 1); Early termination of trial medication (n = 1); Own request (n = 2)) | 16 (Premature visit 3 (n = 5 out of 16): Early study termination (n = 3); Early termination of trial medication (n = 1); Own request (n = 1))
Completed | 16 | 16
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Early study termination | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are reported for all randomized participants, consitent with the intention-to-treat population.
Groups:
- Riociguat: Riociguat Oral Tablet (1 mg, 1.5 mg, 2.0 mg or 2.5 mg three times daily) The dose was individually adjusted in accordance with the in-label titration regimen based on the systemic blood pressure of the patient, the subjects and physicians' subjective estimation and occurrence of adverse reactions. At week 8, the maintenance dose was established and continued for the rest of the study treatment phase
- Placebo: Placebo oral tablet matching riociguat: Sham titration and adjustment to maintenance dose according to individual tolerability as in the experimental arm.
- Total: Total of all reporting groups
Arm/Group | Riociguat | Placebo | Total
Number analyzed (Participants) | 17 | 18 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.18 (7.27) | 65.89 (6.64) | 65.54 (6.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 34
  Male | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 18 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Height [Mean (Standard Deviation); unit: cm] | 161.94 (7.28) | 163.33 (8.14) | 162.66 (7.67)
Weight [Mean (Standard Deviation); unit: kg] | 69.91 (10.9) | 66.84 (11.64) | 68.37 (11.20)
Duration of pulmonary hypertension (PH) [Mean (Standard Deviation); unit: months] | 0.06 (0.24) | 0.56 (1.65) | 0.31 (1.21)
Vital signs - Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] — Population: Systolic blood pressure mesurements of 16 patients in the riociguat arm and 16 patients in the placebo arm were analysed. Values were missing for 2 patients in the placebo arm and one patient in the riociguat arm.
  mmHg
    number analyzed (Participants) | 16 | 16 | 32
    (all) | 132.25 (18.88) | 119.50 (15.27) | 125.88 (18.09)
Vital signs - Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] — Population: Diastolic blood pressure measurements of 16 patients in the riociguat arm and 16 patients in the placebo arm were analysed. Values were missing for 2 patients in the placebo arm and one patient in the riociguat arm.
  mmHg
    number analyzed (Participants) | 16 | 16 | 32
    (all) | 77.13 (9.56) | 73.31 (9.25) | 75.22 (9.45)
Vial signs - Heart rate [Mean (Standard Deviation); unit: beats/min] — Population: Heart rate measurements of 16 patients in the riociguat arm and 16 patients in the placebo arm were analysed. Values were missing for 2 patients in the placebo arm and one patient in the riociguat arm.
  beats/min
    number analyzed (Participants) | 16 | 16 | 32
    (all) | 75.69 (10.13) | 73.44 (8.82) | 74.56 (9.41)
Vital signs - Peripheral Oxygen Saturation (SpO2) [Mean (Standard Deviation); unit: percent] — Population: SpO2 measurements of 16 patients in the riociguat arm and 16 patients in the placebo arm were analysed. Values were missing for 2 patients in the placebo arm and one patient in the riociguat arm.
  percent
    number analyzed (Participants) | 16 | 16 | 32
    (all) | 97.25 (2.05) | 96.56 (1.41) | 96.91 (1.77)
World Health Organization Functional Class (WHO FC) [Count of Participants; unit: Participants] — The World Health Organization (WHO) functional class (FC) describes the severity of pulmonary hypertension (PH) symptoms. FC I is considered the mildest and FC IV the most severe form of PH.
  Participants
    I | 0 | 1 | 1
    II | 16 | 9 | 25
    III | 1 | 8 | 9
    IV | 0 | 0 | 0
Pulmonary hypertension (PH) Etiology [Count of Participants; unit: Participants]
  Idiopathic | 2 | 6 | 8
  Heritable | 0 | 0 | 0
  CTD-associated | 15 | 11 | 26
  other | 0 | 1 | 1
Concomitant diseases [Count of Participants; unit: Participants]
  Treated arterial hypertension | 12 | 8 | 20
  Dyslipidemia | 6 | 5 | 11
  Treated coronary heart disease | 1 | 5 | 6
  Diabetes mellitus | 0 | 2 | 2
  Mild interstitial lung disease | 2 | 7 | 9
  Mild obstructive lung disease | 5 | 3 | 8
  Thyroid dysfunction | 7 | 5 | 12
  Iron deficiency | 5 | 4 | 9
  Oesophagus disease | 4 | 0 | 4
  Degenerative bone disease | 7 | 5 | 12
  Osteoporosis | 2 | 2 | 4
  Autoimmune rheumatic diseases - Systemic Sclerosis (SSc)- limited cutaneous SSc | 6 | 4 | 10
  Autoimmune rheumatic diseases - Systemic Sclerosis (SSc) - diffuse cutaneous SSc | 0 | 1 | 1
  Autoimmune rheumatic diseases - Systemic Sclerosis (SSc) - other subtypes | 6 | 6 | 12
  Autoimmune rheumatic diseases - Sjögren Syndrome | 3 | 1 | 4
  Autoimmune rheumatic diseases - Mixed connective tissue disease | 0 | 2 | 2
  Autoimmune rheumatic diseases - other | 3 | 2 | 5
Blood gas analysis - Saturation of Arterial Oxygen (SaO2) [Mean (Standard Deviation); unit: percent] — Population: SpO2 measurements of 12 patients in the riociguat arm and 14 patients in the placebo arm were analysed. Values were missing for 4 patients in the placebo arm and 5 patients in the riociguat arm.
  percent
    number analyzed (Participants) | 12 | 14 | 26
    (all) | 95.70 (1.20) | 95.97 (1.53) | 95.74 (1.56)
Blood gas analysis - Partial Pressure of Oxygen (PaO2) [Mean (Standard Deviation); unit: mmHg] — Population: PaO2 measurements of 12 patients in the riociguat arm and 14 patients in the placebo arm were analysed. Values were missing for 4 patients in the placebo arm and 5 patients in the riociguat arm.
  mmHg
    number analyzed (Participants) | 12 | 14 | 26
    (all) | 75.57 (9.60) | 79.02 (10.44) | 78.88 (11.14)
Blood gas analysis - Partial Pressure of Carbon Dioxide (PaCO2) [Mean (Standard Deviation); unit: mmHg] — Population: Diastolic blood pressure measurements of 12 patients in the riociguat arm and 14 patients in the placebo arm were analysed. Values were missing for 4 patients in the placebo arm and 5 patients in the riociguat arm.
  mmHg
    number analyzed (Participants) | 14 | 12 | 26
    (all) | 34.09 (4.54) | 36.37 (3.92) | 36.02 (2.92)
Blood gas analysis - pH [Mean (Standard Deviation); unit: pH] — Population: pH measurements of 12 patients in the riociguat arm and 14 patients in the placebo arm were analysed. Values were missing for 4 patients in the placebo arm and 5 patients in the riociguat arm.
  pH
    number analyzed (Participants) | 12 | 14 | 26
    (all) | 7.41 (0.01) | 7.43 (0.02) | 7.42 (0.02)
Blood gas analysis - bicarbonates [Mean (Standard Deviation); unit: mmol/L] — Population: Bicarbonate measurements of 12 patients in the riociguat arm and 14 patients in the placebo arm were analysed. Values were missing for 4 patients in the placebo arm and 5 patients in the riociguat arm
  mmol/L
    number analyzed (Participants) | 12 | 14 | 26
    (all) | 22.34 (1.76) | 24.65 (1.25) | 23.36 (1.64)
Hemodynamics at rest - Right Arterial Pressure (RAP) [Mean (Standard Deviation); unit: mmHg] | 6.71 (3.12) | 5.28 (2.85) | 5.97 (3.02)
Hemodynamics at rest - Systolic Pulmonary Artery Pressure (sPAP) [Mean (Standard Deviation); unit: mmHg] | 36.88 (4.33) | 36.61 (3.85) | 36.74 (4.03)
Hemodynamics at rest - diastolic pulmonary artery pressure (dPAP) [Mean (Standard Deviation); unit: mmHg] | 15.47 (1.94) | 14.44 (2.25) | 14.94 (2.14)
Hemodynamics at rest - mean pulmonary arterial pressure (mPAP) [Mean (Standard Deviation); unit: mmHg] | 24.06 (2.56) | 23.67 (2.87) | 23.86 (2.69)
Hemodynamics at rest - pulmonary artery wedge pressure (PAWP) [Mean (Standard Deviation); unit: mmHg] | 9.83 (3.59) | 10.18 (2.27) | 10.00 (2.98)
Hemodynamics at rest - cardiac output (CO) [Mean (Standard Deviation); unit: l/min] | 4.62 (0.93) | 4.70 (1.06) | 4.66 (0.99)
Hemodynamics at rest - cardiac index (CI) [Mean (Standard Deviation); unit: l/min/m2] | 2.70 (0.43) | 2.74 (0.64) | 2.72 (0.51)
Hemodynamics at rest - Pulmonary Vascular Resistance (PVR) [Mean (Standard Deviation); unit: WU] | 3.09 (0.85) | 2.93 (0.59) | 3.01 (0.73)
Hemodynamics at rest - Venous Oxygen Saturation (SVO2) [Mean (Standard Deviation); unit: percent] | 72.53 (11.24) | 59.89 (5.9) | 71.17 (8.87)
Six-minute walking distance (6MWD) test - 6MWD [Mean (Standard Deviation); unit: m] — Population: 6MWD of 16 patients in the riociguat arm and 18 patients in the placebo arm was analysed. Values were missing for 1 patient in the riociguat arm.
  m
    number analyzed (Participants) | 16 | 18 | 34
    (all) | 431.13 (53.24) | 387.11 (81.94) | 407.82 (72.42)
Six-minute walking distance (6MWD) test - Peripheral Oxygen Saturation (SpO2) (test end) [Mean (Standard Deviation); unit: percent] — Population: 6MWD of 16 patients in the riociguat arm and 18 patients in the placebo arm was analysed. Values were missing for 1 patient in the riociguat arm.
  percent
    number analyzed (Participants) | 16 | 18 | 34
    (all) | 87.94 (9.22) | 89.39 (11.61) | 88.71 (10.42)
Six-minute walking distance (6MWD) test - Borg dyspnea score [Mean (Standard Deviation); unit: scores on a scale] — The Borg Scale (Breathlessness Scale) is commonly used to measure shortness of breath of patients or in sports medicine. In this study, the Borg Scale was applied to record dyspnea immediately following the 6-minute walk test.
  The Borg Scale according to the ATS guidelines (ATS 2002) ranges from 0 (no dyspnea at all) to 10 (maximal dyspnea) Population: 6MWD of 16 patients in the riociguat arm and 18 patients in the placebo arm was analysed. Values were missing for 1 patient in the riociguat arm.
  scores on a scale
    number analyzed (Participants) | 16 | 18 | 34
    (all) | 3.53 (2.35) | 2.69 (1.83) | 3.09 (2.10)
Short Form-36 Health Survey - Physical functioning [Mean (Standard Deviation); unit: scores on a scale] — Quality of Life (QoL) was assessed using the SF 36-questionnaire. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale, i.e. a score of 0 is equivalent to maximum disability and a score of 100 is equivalent to no disability.
  Sections: vitality; physical functioning; bodily pain; general health perceptions; physical role functioning; emotional role functioning; social role functioning; mental health. Two summation scores, physical and mental summation score, were calculated. Population: The SF-36 survey of 16 patients in the riociguat arm and 18 patients in the placebo arm was analysed. Values were missing for 1 patient in the riociguat arm.
  scores on a scale
    number analyzed (Participants) | 16 | 18 | 34
    (all) | 59.38 (23.66) | 59.17 (23.28) | 59.26 (23.10)
Short Form-36 Health Survey - Physical role function [Mean (Standard Deviation); unit: scores on a scale] — Quality of Life (QoL) was assessed using the SF 36-questionnaire. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale, i.e. a score of 0 is equivalent to maximum disability and a score of 100 is equivalent to no disability.
  Sections: vitality; physical functioning; bodily pain; general health perceptions; physical role functioning; emotional role functioning; social role functioning; mental health. Two summation scores, physical and mental summation score, were calculated. Population: The SF-36 survey of 16 patients in the riociguat arm and 18 patients in the placebo arm was analysed. Values were missing for 1 patient in the riociguat arm.
  scores on a scale
    number analyzed (Participants) | 16 | 18 | 34
    (all) | 48.44 (41.30) | 31.94 (56.10) | 39.71 (46.66)
Short Form-36 Health Survey - Pain [Mean (Standard Deviation); unit: scores on a scale] — Quality of Life (QoL) was assessed using the SF 36-questionnaire. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale, i.e. a score of 0 is equivalent to maximum disability and a score of 100 is equivalent to no disability.
  Sections: vitality; physical functioning; bodily pain; general health perceptions; physical role functioning; emotional role functioning; social role functioning; mental health. Two summation scores, physical and mental summation score, were calculated Population: The SF-36 survey of 16 patients in the riociguat arm and 18 patients in the placebo arm was analysed. Values were missing for 1 patient in the riociguat arm.
  scores on a scale
    number analyzed (Participants) | 16 | 18 | 34
    (all) | 63.56 (25.81) | 62.78 (20.83) | 63.15 (22.94)
Short Form-36 Health Survey - General health perception [Mean (Standard Deviation); unit: scores on a scale] — Quality of Life (QoL) was assessed using the SF 36-questionnaire. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale, i.e. a score of 0 is equivalent to maximum disability and a score of 100 is equivalent to no disability.
  Sections: vitality; physical functioning; bodily pain; general health perceptions; physical role functioning; emotional role functioning; social role functioning; mental health. Two summation scores, physical and mental summation score, were calculated Population: The SF-36 survey of 16 patients in the riociguat arm and 18 patients in the placebo arm was analysed. Values were missing for 1 patient in the riociguat arm.
  scores on a scale
    number analyzed (Participants) | 16 | 18 | 34
    (all) | 51.88 (14.89) | 53.06 (23.67) | 52.50 (19.74)
Short Form-36 Health Survey - Vitality [Mean (Standard Deviation); unit: scores on a scale] — Quality of Life (QoL) was assessed using the SF 36-questionnaire. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale, i.e. a score of 0 is equivalent to maximum disability and a score of 100 is equivalent to no disability.
  Sections: vitality; physical functioning; bodily pain; general health perceptions; physical role functioning; emotional role functioning; social role functioning; mental health. Two summation scores, physical and mental summation score, were calculated Population: The SF-36 survey of 16 patients in the riociguat arm and 18 patients in the placebo arm was analysed. Values were missing for 1 patient in the riociguat arm.
  scores on a scale
    number analyzed (Participants) | 16 | 18 | 34
    (all) | 40.31 (19.01) | 46.11 (17.62) | 43.38 (18.25)
Short Form-36 Health Survey - Social functioning [Mean (Standard Deviation); unit: scores on a scale] — Quality of Life (QoL) was assessed using the SF 36-questionnaire. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale, i.e. a score of 0 is equivalent to maximum disability and a score of 100 is equivalent to no disability.
  Sections: vitality; physical functioning; bodily pain; general health perceptions; physical role functioning; emotional role functioning; social role functioning; mental health. Two summation scores, physical and mental summation score, were calculated Population: The SF-36 survey of 16 patients in the riociguat arm and 18 patients in the placebo arm was analysed. Values were missing for 1 patient in the riociguat arm.
  scores on a scale
    number analyzed (Participants) | 16 | 18 | 34
    (all) | 65.06 (26.59) | 72.39 (22.05) | 68.94 (24.20)
Short Form-36 Health Survey - Emotional role function [Mean (Standard Deviation); unit: scores on a scale] — Quality of Life (QoL) was assessed using the SF 36-questionnaire. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale, i.e. a score of 0 is equivalent to maximum disability and a score of 100 is equivalent to no disability.
  Sections: vitality; physical functioning; bodily pain; general health perceptions; physical role functioning; emotional role functioning; social role functioning; mental health. Two summation scores, physical and mental summation score, were calculated Population: The SF-36 survey of 16 patients in the riociguat arm and 18 patients in the placebo arm was analysed. Values were missing for 1 patient in the riociguat arm.
  scores on a scale
    number analyzed (Participants) | 16 | 18 | 34
    (all) | 47.94 (47.12) | 38.89 (53.97) | 43.15 (50.30)
Short Form-36 Health Survey - Mental well-being [Mean (Standard Deviation); unit: scores on a scale] — Quality of Life (QoL) was assessed using the SF 36-questionnaire. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale, i.e. a score of 0 is equivalent to maximum disability and a score of 100 is equivalent to no disability.
  Sections: vitality; physical functioning; bodily pain; general health perceptions; physical role functioning; emotional role functioning; social role functioning; mental health. Two summation scores, physical and mental summation score, were calculated Population: The SF-36 survey of 16 patients in the riociguat arm and 18 patients in the placebo arm was analysed. Values were missing for 1 patient in the riociguat arm.
  scores on a scale
    number analyzed (Participants) | 16 | 18 | 34
    (all) | 63.50 (17.64) | 65.33 (15.70) | 64.47 (16.41)
Short Form-36 Health Survey - Physical summation score [Mean (Standard Deviation); unit: scores on a scale] — Quality of Life (QoL) was assessed using the SF 36-questionnaire. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale, i.e. a score of 0 is equivalent to maximum disability and a score of 100 is equivalent to no disability.
  Sections: vitality; physical functioning; bodily pain; general health perceptions; physical role functioning; emotional role functioning; social role functioning; mental health. Two summation scores, physical and mental summation score, were calculated Population: The SF-36 survey of 16 patients in the riociguat arm and 18 patients in the placebo arm was analysed. Values were missing for 1 patient in the riociguat arm.
  scores on a scale
    number analyzed (Participants) | 16 | 18 | 34
    (all) | 52.50 (20.19) | 50.56 (23.36) | 51.47 (21.62)
Short Form-36 Health Survey - Mental summation score [Mean (Standard Deviation); unit: scores on a scale] — Quality of Life (QoL) was assessed using the SF 36-questionnaire. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale, i.e. a score of 0 is equivalent to maximum disability and a score of 100 is equivalent to no disability.
  Sections: vitality; physical functioning; bodily pain; general health perceptions; physical role functioning; emotional role functioning; social role functioning; mental health. Two summation scores, physical and mental summation score, were calculated Population: The SF-36 survey of 16 patients in the riociguat arm and 18 patients in the placebo arm was analysed. Values were missing for 1 patient in the riociguat arm.
  scores on a scale
    number analyzed (Participants) | 16 | 18 | 34
    (all) | 53.75 (18.92) | 55.22 (19.44) | 54.53 (18.92)
Echocardiography at rest - Estimated Systolic Pulmonary Artery Pressure (sPAP) [Mean (Standard Deviation); unit: mmHg] — Population: sPAP estimates of 17 patients in the riociguat arm and 16 patients in the placebo arm was analysed. Values were missing for 2 patients in the placebo arm.
  mmHg
    number analyzed (Participants) | 17 | 16 | 33
    (all) | 35.06 (7.58) | 31.94 (7.34) | 33.55 (7.52)
Echocardiography at rest - right atrial (RA) area [Mean (Standard Deviation); unit: cm2] | 12.47 (3.04) | 13.56 (2.66) | 13.03 (2.86)
Echocardiography at rest - right ventricular (RV) area [Mean (Standard Deviation); unit: cm2] — Population: RV area measurements of 15 patients in the riociguat arm and 14 patients in the placebo arm were analysed. Values were missing for 4 patients in the placebo arm and for 2 patients in the riociguat arm.
  cm2
    number analyzed (Participants) | 15 | 14 | 29
    (all) | 12.53 (2.85) | 13.64 (2.65) | 13.07 (2.76)
Echocardiography at rest - Tricuspid Annular Plane Systolic Excursion (TAPSE) [Mean (Standard Deviation); unit: cm] | 2.37 (0.41) | 2.30 (0.48) | 2.33 (0.44)
Echocardiography at rest - left ventricular eccentricity index (LV-EI) [Mean (Standard Deviation); unit: index] — LV-EI is the ratio of septical-parallel to septical-perdendicular left ventricular diameters in parasternal short-axis view; normal = 1, increased (≥ 1.1) indicates right ventricular pressure/volume overload Population: LV-EI of 15 patients in the riociguat arm and 14 patients in the placebo arm was analysed. Values were missing for 6 patients in the placebo arm and for 3 patients in the riociguat arm.
  index
    number analyzed (Participants) | 14 | 12 | 26
    (all) | 1.64 (2.41) | 1.00 (0.00) | 1.35 (1.77)
Echocardiography at rest - Left ventricular ejection fraction [Mean (Standard Deviation); unit: percent] | 62.82 (6.65) | 65.28 (5.84) | 64.09 (6.28)
Lung function - Forced Vital Capacity (FVC) [Mean (Standard Deviation); unit: L] — Population: FVC measurements of 12 patients in the riociguat arm and 13 patients in the placebo arm were analysed. Values were missing for 5 patients in the placebo arm and for 5 patients in the riociguat arm.
  L
    number analyzed (Participants) | 12 | 13 | 25
    (all) | 92.18 (12.54) | 88.80 (16.22) | 90.42 (14.37)
Lung function - Forced expiratory volume in the first second (FEV1) [Mean (Standard Deviation); unit: percent predicted] — Population: FEV1 measurements of 12 patients in the riociguat arm and 13 patients in the placebo arm were analysed. Values were missing for 5 patients in the placebo arm and for 5 patients in the riociguat arm.
  percent predicted
    number analyzed (Participants) | 12 | 13 | 25
    (all) | 93.87 (14.80) | 90.90 (15.74) | 92.32 (15.05)
Lung function - total lung capacity (TLC) [Mean (Standard Deviation); unit: percent (predicted)] — Population: TLC measurements of 12 patients in the riociguat arm and 11 patients in the placebo arm were analysed. Values were missing for 7 patients in the placebo arm and for 5 patients in the riociguat arm.
  percent (predicted)
    number analyzed (Participants) | 12 | 11 | 23
    (all) | 96.71 (11.68) | 87.45 (11.97) | 92.28 (12.48)
Lung function - Residual volume [Mean (Standard Deviation); unit: percent predicted] — Population: Residual Volume measurements of 12 patients in the riociguat arm and 11 patients in the placebo arm were analysed. Values were missing for 7 patients in the placebo arm and for 5 patients in the riociguat arm.
  percent predicted
    number analyzed (Participants) | 11 | 12 | 23
    (all) | 99.48 (30.41) | 88.54 (21.67) | 94.25 (26.59)
Lung function - Diffusion limited carbon monoxide (DLCO) [Mean (Standard Deviation); unit: percent predicted] — diffusing capacity of the lung Population: DLCO measurements of 11 patients in the riociguat arm and 13 patients in the placebo arm were analysed. Values were missing for 5 patients in the placebo arm and for 6 patients in the riociguat arm.
  percent predicted
    number analyzed (Participants) | 13 | 11 | 24
    (all) | 62.15 (12.47) | 56.01 (7.00) | 58.83 (10.15)
Lung function - Diffusion limited carbon monoxide/alevolar volume (DLCO/VA) [Mean (Standard Deviation); unit: percent predicted] — diffusing capacity normalized to alveolar volume Population: DLCO/VA of 2 patients in the riociguat arm and 5 patients in the placebo arm were analysed. Values were missing for 13 patients in the placebo arm and for 15 patients in the riociguat arm.
  percent predicted
    number analyzed (Participants) | 2 | 5 | 7
    (all) | 67.15 (10.25) | 72.52 (17.51) | 70.99 (15.12)
Laboratory - Hemoglobin [Mean (Standard Deviation); unit: g/dl] — Population: Hemoglobin measurements of 12 patients in the riociguat arm and 15 patients in the placebo arm were analysed. Values were missing for 3 patients in the placebo arm and for 5 patients in the riociguat arm.
  g/dl
    number analyzed (Participants) | 12 | 15 | 27
    (all) | 13.23 (1.81) | 13.29 (0.71) | 13.26 (1.29)
Laboratory - Creatinine [Mean (Standard Deviation); unit: mg/dl] — Population: Creatinine measurements of 12 patients in the riociguat arm and 15 patients in the placebo arm were analysed. Values were missing for 3 patients in the placebo arm and for 5 patients in the riociguat arm.
  mg/dl
    number analyzed (Participants) | 12 | 15 | 27
    (all) | 0.73 (0.15) | 0.84 (0.24) | 0.79 (0.21)
Laboratory - Urea [Mean (Standard Deviation); unit: mg/dl] — Population: Urea measurements of 11 patients in the riociguat arm and 15 patients in the placebo arm were analysed. Values were missing for 3 patients in the placebo arm and for 6 patients in the riociguat arm.
  mg/dl
    number analyzed (Participants) | 11 | 15 | 26
    (all) | 25.82 (6.68) | 30.53 (14.61) | 28.54 (11.96)
Laboratory - Uric acid [Mean (Standard Deviation); unit: mg/dl] — Population: Uric acid measurements of 11 patients in the riociguat arm and 14 patients in the placebo arm were analysed. Values were missing for 4 patients in the placebo arm and for 6 patients in the riociguat arm.
  mg/dl
    number analyzed (Participants) | 11 | 14 | 25
    (all) | 4.49 (0.81) | 4.93 (2.10) | 4.74 (1.65)
Laboratory - Serum Glutamic Pyruvic Transaminase (SGPT) [Mean (Standard Deviation); unit: U/L] — Population: SGPT measurements of 12 patients in the riociguat arm and 15 patients in the placebo arm were analysed. Values were missing for 3 patients in the placebo arm and for 5 patients in the riociguat arm.
  U/L
    number analyzed (Participants) | 12 | 15 | 27
    (all) | 18.25 (15.22) | 22.27 (13.74) | 20.48 (14.28)
Laboratory - C-reactive protein (CRP) [Mean (Standard Deviation); unit: mg/L] — Population: CRP measurements of 12 patients in the riociguat arm and 14 patients in the placebo arm were analysed. Values were missing for 4 patients in the placebo arm and for 5 patients in the riociguat arm.
  mg/L
    number analyzed (Participants) | 12 | 14 | 26
    (all) | 3.27 (2.23) | 6.15 (8.50) | 4.82 (6.48)
Laboratory - N-terminal prohormone of brain natriuretic peptide (NTproBNP) [Mean (Standard Deviation); unit: pg/ml] — Population: NTproBNP measurements of 12 patients in the riociguat arm and 15 patients in the placebo arm were analysed. Values were missing for 3 patients in the placebo arm and for 5 patients in the riociguat arm.
  pg/ml
    number analyzed (Participants) | 12 | 15 | 27
    (all) | 331.08 (361.44) | 316.73 (342.13) | 323.11 (344.02)

OUTCOME MEASURES:

1. Primary Outcome: Change of Pulmonary Vascular Resistance (PVR)
Description: Change in pulmonary hemodynamics assessed by right heart catheterization
Time Frame: baseline, 24 weeks
Population: All randomized participants were included in the analysis (intention-to-treat population). The number of analyzed paticipants may vary due to missing data for specific outcome measures. The per-protocol set is identical to the intention-to-treat set, as no major protocol deviations occurred and all participants met the predefined eligibility criteria.
Measure: Mean (Standard Deviation); unit: WU
Groups:
- Riociguat: Riociguat Oral Tablet: Riociguat Oral Tablet (1 mg, 1.5 mg, 2.0 mg or 2.5 mg three times daily): individually adjusted dose in accordance with the in-label titration regimen (maximum dosage of 2.5mg tid). At week 8, the maintenance dose was established and maintained for the rest of study participation.
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 14 | 15
WU | -0.69 (0.60) | 0.89 (3.29)
Statistical Analysis 1: Comparison: Riociguat vs Placebo; Test type: Superiority; p = 0.043, ANCOVA; baseline value as covariate
Statistical Analysis 2: Comparison: Riociguat vs Placebo; Test type: Other — Sensitivity analysis; p = 0.045, Multiple imputation

2. Secondary Outcome: Change of Cardiac Index (CI) at Rest From Baseline at 24 Weeks
Description: Change in pulmonary hemodynamics assessed by right heart catheterization
Time Frame: baseline, 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: l/min/m2
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 14 | 15
l/min/m2 | 0.21 (0.54) | -0.07 (0.40)
Statistical Analysis 1: Comparison: Riociguat vs Placebo; Secondary endpoints statistically analyzed by a hierarchical testing strategy; Test type: Superiority; p = 0.116, t-test, 2 sided; Mean Difference (Final Values) = -0.28, 95% CI 2-sided [-0.64 to 0.08]

3. Secondary Outcome: Change of Total Pulmonary Resistance (TPR) From Baseline at 24 Weeks
Description: Change in Pulmonary hemodynamics assessed by right heart catheterization
  Hierarchical testing of secondary endpoints stopped after first step.
Time Frame: baseline, 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg·min/L
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 14 | 15
mmHg·min/L | 0.51 (1.18) | -0.21 (0.82)

4. Secondary Outcome: Change of Diffusion Capacity of the Lung (DLCO) From Baseline at 24 Weeks
Description: Change assessed by lung function tests.
  Hierarchical testing of secondary endpoints stopped after first step.
Time Frame: baseline, 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent predicted
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 11 | 13
percent predicted | 1.16 (6.40) | 0.09 (7.40)

5. Secondary Outcome: Change in 6-minute Walking Distance (6MWD)
Description: Change in exercise capacity assessed by 6-minute walking distance test
  Hierarchical testing of secondary endpoints stopped after first step.
Time Frame: baseline, 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: m
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 16 | 16
m | 23 (56.41) | 24 (43.58)

6. Secondary Outcome: Change of World Health Organization- Functional Class (WHO-FC) From Baseline at 24 Weeks
Description: Change of WHO functional class, change score The World Health Organization (WHO) functional class (FC) describes the severity of pulmonary hypertension (PH) symptoms. FC I is considered the mildest and FC IV the most severe form of PH.
Time Frame: baseline, 24 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 16 | 16
Participants
  Improvement | 2 | 3
  Worsening | 0 | 1
  Unchanged | 14 | 12

7. Other Pre Specified Outcome: Change of World Health Organization- Functional Class (WHO-FC) From Baseline at 12 Weeks
Description: as for outcome 6
Time Frame: baseline, 12 weeks
Population: All randomized participants were included in the analysis (intention-to-treat population). The number of analyzed paticipants may vary due to missing data for specific outcome measures.
Measure: Count of Participants; unit: Participants
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 13 | 14
Participants
  Improvement (-1) | 0 | 3
  Worsening (+1) | 1 | 0
  Unchanged | 12 | 11

8. Other Pre Specified Outcome: Change in Quality of Life (QoL) From Baseline at 24 Weeks
Description: Quality of Life (QoL) was assessed using the Short Form (SF) 36-questionnaire. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale, i.e. a score of 0 is equivalent to maximum disability and a score of 100 is equivalent to no disability.
  Sections: vitality; physical functioning; bodily pain; general health perceptions; physical role functioning; emotional role functioning; social role functioning; mental health. Two summation scores, physical and mental summation score, were calculated
Time Frame: baseline, 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 15 | 15
scores on a scale
  Physical functioning | 4.00 (15.38) | 2.00 (21.61)
  Physical role function | -5.00 (34.33) | 31.67 (53.00)
  Pain | -1.33 (19.35) | 9.53 (22.51)
  General health perception | -5.13 (13.67) | 0.60 (15.37)
  Vitality | -1.67 (14.47) | 5.33 (16.09)
  Social functioning | 1.73 (23.88) | 6.67 (14.78)
  Emotional role function | 15.53 (48.59) | 40.13 (58.02)
  Mental well-being | 2.40 (12.36) | 4.53 (7.84)
  Physical summation score | -1.67 (11.89) | 9.73 (18.39)
  Mental summation score | 2.60 (16.97) | 11.33 (14.32)

9. Other Pre Specified Outcome: Change in Forced Expiratory Volume in 1 Second (FEV1) From Baseline at 24 Weeks
Description: Lung function and lung diffusing capacity
Time Frame: baseline, 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent predicted
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 3 | 5
percent predicted | 0.37 (2.09) | 1.04 (5.99)

10. Other Pre Specified Outcome: Change in Total Lung Capacity (TLC) From Baseline at 24 Weeks
Description: Lung function and lung diffusing capacity
Time Frame: baseline, 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent predicted
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 12 | 11
percent predicted | -4.70 (12.66) | -0.91 (8.78)

11. Other Pre Specified Outcome: Change in Diffusing Capacity of the Lung (DLCO)
Description: Lung function and lung diffusing capacity
Time Frame: baseline, 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent predicted
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 11 | 13
percent predicted | 0.09 (7.40) | 1.16 (6.40)

12. Other Pre Specified Outcome: Change in Systolic Pulmonary Arterial Pressure (sPAP) From Baseline at 24 Weeks
Description: Change in systolic pulmonary arterial pressure (sPAP) from baseline at 24 weeks assessed by echocardiography
Time Frame: baseline, 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 15 | 12
mmHg | -5.20 (7.26) | -3.42 (7.06)

13. Other Pre Specified Outcome: Change in Right Ventricular Area (RV-area) From Baseline at 24 Weeks
Description: Change in right ventricular area (RV-area) from baseline at 24 weeks assessed by echocardiography
Time Frame: baseline, 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm2
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 15 | 12
cm2 | 0.00 (2.51) | -1.33 (1.97)

14. Other Pre Specified Outcome: Change in Right Atrial Area (RA-area) From Baseline at 24 Weeks
Description: Change in right atrial area (RA-area) from baseline at 24 weeks assessed by echocardiography
Time Frame: baseline, 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm2
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 16 | 16
cm2 | 0.38 (3.34) | -0.68 (2.27)

15. Other Pre Specified Outcome: Change in Tricuspid Annular Plane Systolic Excursion (TAPSE) From Baseline at 24 Weeks
Description: Change in tricuspid annular plane systolic excursion (TAPSE) from baseline at 24 weeks assessed by echocardiography
Time Frame: baseline, 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 16 | 16
cm | 0.15 (0.34) | -0.08 (0.58)

16. Other Pre Specified Outcome: Change in Left Ventricular Eccentricity Index (LV-EI) From Baseline at 24 Weeks
Description: Change in left ventricular eccentricity index (LV-EI) from baseline at 24 weeks assessed by echocardiography.
  LV-EI is the ratio of septical-parallel to septical-perdendicular left ventricular diameters in parasternal short-axis view; normal = 1, increased (≥ 1.1) indicates right ventricular pressure/volume overload
Time Frame: baseline, 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 14 | 12
index | -0.62 (2.41) | 0.00 (0.12)

17. Other Pre Specified Outcome: Change in N-terminal Prohormone of Brain Natriuretic Peptide (NT-pro BNP) From Baseline at 12 Weeks
Description: blood analysis
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 9 | 11
pg/ml | -116,3333 (229,11951) | -8,7273 (212,47545)

18. Other Pre Specified Outcome: Change in N-terminal Prohormone of Brain Natriuretic Peptide (NT-pro BNP) From Baseline at 24 Weeks
Description: blood analysis
Time Frame: baseline, 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 12 | 14
pg/ml | -86.50 (246.40) | -4.57 (251.30)

19. Other Pre Specified Outcome: Change in Oxygen Partial Pressure (PaO2) From Baseline at 24 Weeks
Description: Change in oxygen partial pressure (PaO2) from baseline at 24 weeks assessed by blood gas analysis
Time Frame: baseline, 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 12 | 13
mmHg | -2.83 (7.99) | -3.38 (12.22)

20. Other Pre Specified Outcome: Change in Carbon Dioxide Partial Pressure (PCO2)
Description: blood gas analysis
Time Frame: baseline, 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 12 | 13
mmHg | 0.48 (2.73) | -0.83 (3.75)

21. Other Pre Specified Outcome: Change Oxygen Saturation of the Blood (SaO2)
Description: Change oxygen saturation of the blood (SaO2) assessed by blood gas analysis
Time Frame: baseline, 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent SaO2
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 12 | 12
percent SaO2 | -0.36 (1.08) | -0.87 (3.58)

22. Other Pre Specified Outcome: Change in pH
Description: blood gas analysis
Time Frame: baseline,24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 12 | 13
pH | 0.01 (0.03) | 0.00 (0.03)

23. Other Pre Specified Outcome: Change in Bicarbonates
Description: blood gas analysis
Time Frame: baseline, 24 weeks
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 12 | 13
mmol/L | 0.80 (1.63) | -0.43 (1.44)

24. Other Pre Specified Outcome: Change in Base Excess
Description: Change in base excess assessed by blood gas analysis
Time Frame: baseline, 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 12 | 13
mmol/L | 0.74 (1.63) | -0.34 (1.46)

25. Other Pre Specified Outcome: Change in Systolic Pulmonary Arterial Pressure (sPAP)
Description: Pulmonary hemodynamics assessed by right heart catheterization
Time Frame: baseline, 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 14 | 15
mmHg | -2.36 (6.22) | -3.00 (5.72)

26. Other Pre Specified Outcome: Change in Mean Pulmonary Arterial Pressure (mPAP)
Description: Pulmonary hemodynamics assessed by right heart catheterization
Time Frame: baseline, 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 14 | 15
mmHg | -1.43 (5.2) | -1.60 (4.39)

27. Other Pre Specified Outcome: Change in dPAP (Diastolic Pulmonary Artery Pressure)
Description: Pulmonary hemodynamics assessed by right heart catheterization
Time Frame: baseline, 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 14 | 15
mmHg | -1.43 (3.16) | -0.27 (4.43)

28. Other Pre Specified Outcome: Change in PAWP (Pulmonary Artery Wedge Pressure)
Description: Pulmonary hemodynamics assessed by right heart catheterization
Time Frame: baseline, 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 14 | 15
mmHg | 1.36 (2.95) | -0.53 (3.14)

29. Other Pre Specified Outcome: Change in RAP (Right Atrial Pressure)
Description: Pulmonary hemodynamics assessed by right heart catheterization
Time Frame: baseline, 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 14 | 15
mmHg | 0.5 (2.44) | 0.33 (2.74)

30. Other Pre Specified Outcome: Change in Cardiac Output and Ejection Fraction (CO)
Description: Pulmonary hemodynamics assessed by right heart catheterization
Time Frame: baseline, 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 14 | 15
L/min | 0.35 (0.86) | -0.19 (0.75)

31. Other Pre Specified Outcome: Change in Central Venous Saturation (SvO2)
Description: blood gas analysis
Time Frame: baseline, 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent SvO2
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 14 | 15
percent SvO2 | 1.07 (11.02) | 3.20 (5.45)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from baseline until safety follow-up (30 ± 14 days after last intake of study drug). With a treatment phase of 24 weeks (± 14 days), the overall adverse event data collection period corresponds to approximately 28 weeks.
Arm/Group | Riociguat | Placebo
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/18
Serious Adverse Events (participants affected / at risk) | 2/17 | 1/18
Other Adverse Events (participants affected / at risk) | 16/17 | 16/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Riociguat (N=17) | Placebo (N=18)
Bradycardia (Cardiac disorders) | 1 | 0
Gastrointestinal bleeding (Gastrointestinal disorders) | 1 | 0
Knee endoprothesis (Surgical and medical procedures) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Commotio cerebri (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Riociguat (N=17) | Placebo (N=18)
Nausea (Gastrointestinal disorders) | 5 | 4
Bloating (Gastrointestinal disorders) | 0 | 2
Emesis (Gastrointestinal disorders) | 2 | 2
Diarrhea (Gastrointestinal disorders) | 3 | 2
Flatulence (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 2
Gastritis (Gastrointestinal disorders) | 1 | 3
Reflux (Gastrointestinal disorders) | 5 | 2
Pain (Musculoskeletal and connective tissue disorders) | 4 | 4
Headache (Musculoskeletal and connective tissue disorders) | 6 | 5
Fatigue (Musculoskeletal and connective tissue disorders) | 1 | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Infections (any) (Respiratory, thoracic and mediastinal disorders) | 9 | 5
COVID-19 (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Hypotension (Cardiac disorders) | 4 | 3
Dizziness (Cardiac disorders) | 3 | 7
Edema (Cardiac disorders) | 1 | 2
Chest pain (Cardiac disorders) | 2 | 0
Palpitations (Cardiac disorders) | 5 | 6
Urinary tract infection (Renal and urinary disorders) | 1 | 1
Night sweats (General disorders) | 2 | 0

LIMITATIONS AND CAVEATS:
Sample size reduction to 50% limits statistical power in this two-armed study design. 24-week treatment may have been too short to assess long-term outcomes, especially with reduced exposure due to early end of study (not safety-related). Drug effects may appear less distinct (verum), clinical worsening less pronounced (control), reducing effect size. Baseline imbalances and placebo effects affected interpretation of subjective endpoints. No advanced imaging/biomarker endpoints were included.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has first publication rights, intended to be a joint, multi-center publication.

Subsequent publications by Institution and/or Investigator require at least 60-day sponsor review. Sponsor may remove any information considered confidential and/or proprietary or would hinder the marketing authorization holder in the further development of the Investigational Product. Sponsor may request changes or delay (max 180 days) if patentability is affected. Scientific neutrality must be preserved.

DOCUMENTS (2):
  • Study Protocol (2025-01-15): https://cdn.clinicaltrials.gov/large-docs/87/NCT05339087/Prot_000.pdf
  • Statistical Analysis Plan (2025-08-07): https://cdn.clinicaltrials.gov/large-docs/87/NCT05339087/SAP_001.pdf